CLINICAL TRIAL: NCT02904252
Title: The Prevalence and Severity of HCV Infection in Thalassemia Major and Thalassemia Intermedia in Siriraj Hospital
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 481/2558
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C; Fibrosis; Thalassemia
Keywords: Transient elastography; Fibrotest
MeSH Terms: conditions — Hepatitis C; Fibrosis; Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Clotted blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Population : The participants are thalassemia patients who regularly visit Hematology Clinic, Department of Medicine, Faculty of Medicine Siriraj Hospital Clinical data, Laboratory data (Blood samples) and Transient elastography data will be collected from all participants, as previously described.
  Interventions: Other: Transient elastography

INTERVENTIONS:
Other: Transient elastography — Transient elastography (TE) is an ultrasound-based device used for measuring the degree of liver stiffness. A transducer probe is used to create mild amplitude and low frequency vibrations (50 Hz) that transmitted through the liver tissue. This results in an elastic shear wave that propagates through the underlying liver tissue. The probe then utilizes pulse-echo ultrasound to follow the propagation of the shear wave and to measure its velocity. The velocity of the wave is directly related to tissue stiffness which correlates with fibrosis. The sensitivity and the specificity of TE is between 68%-88% and between 66%-100%, respectively for the detection of significant liver fibrosis (METAVIR score F>2).
  Other Names: Fibroscan

SUMMARY:
The primary objective is to assess the prevalence and genotypes of HCV infection in thalassemia major and thalassemia intermediate patients who have received blood transfusion in the Department of Medicine, Faculty of Medicine Siriraj Hospital.

The secondary objective is to identify the effect of HCV infection as well as the risk factors of advanced liver disease and liver cirrhosis in these patients

The third objective is to identify the role of serum HA level and fibrotest in the prediction of cirrhosis in these patients.

DETAILED DESCRIPTION:
Study protocol

Data collection:

The eligible patients will be asked to participate in the study. After signing informed consent, the patients will be asked to complete questionnaire, all clinical and laboratory data of the patients will be retrieved from out-patient electronic or paper medical records, electronic laboratory results. The data will include the followings:

1. Clinical data

   * Demographic information (age, gender, ethnicity, education, marital status)
   * Family history of liver disease
   * Current relevant medication
   * Weight, height and body mass index (BMI) at the time of enrollment
   * History of blood or blood product transfusion, last transfusion
   * History of alcohol consumption
   * History of active liver disease
2. Laboratory data

   * Complete blood count
   * Iron study (serum ferritin, serum iron, total iron binding capacity and transferrin saturation)
   * Hemoglobin typing
   * HIV antibody status (only if available)
   * liver biochemistry including AST, ALT, albumin, globulin
   * Blood urea nitrogen, creatinine
   * HBsAg, Anti-HBsAb
   * Anti-HCV antibody
   * HCV RNA, HCV genotyping (only in patients with positive Anti-HCV)
   * Serum hyaluronic acid
   * Fibrotest

After data collection, all patients will receive blood test for serum hyaluronic acid. If the patients have incomplete laboratory data (except HIV antibody status), they will receive additional blood tests for missing data. All patients will be appointed for transient elastography. All the cost for the extra-investigation will be supported by the study.

Transient elastography (TE or Fibroscan):

TE will be used to evaluate liver fibrosis. TE will be performed in all patients by examiners who were blind to clinical, laboratory data. The right lobe of the liver was targeted through an intercostal space access while the patient was lying in the dorsal decubitus position with the right arm in maximal abduction. With the assistance of TE, a liver portion of at least 6-cm thickness, free of large vessels, was identified for examination. The rate of successful measurements was interpreted by the ratio between the number of those validated and total number of measurements. The results were expressed as a median value of the total measurements in kPa. Patients with ascites were excluded from the study due to the limitation of result interpretation.

Data Handling :

Data of each patient will be collected at the OPD, Division of Hematology and Division of Gastroenterology, Siriraj Hospital, Mahidol University, Bangkok, Thailand.

The study will be started after it is approved by the Ethics Committee ofSiriraj Hospital. Patients' identification number will be stored in a separate log book. Results will be reported at the aggregate level only, and individual-level data will never be released.

Sample Size and Statistical analysis Sample size The primary research question of this study is to assess the prevalence of HCV infection in thalassemia major and thalassemia intermediate patients who received prior blood transfusion. From the previous research conducted by Wanachiwanawin W, et al , we estimate that the prevalence of hepatitis C viral infection in thalassemia patient is 20 percent. The sample size is 246 samples according to the calculation with 95 % confident interval.

Statistical analysis

1. The quantitative data, such as age, will be analyzed by mean and standard deviation or by mode and median (in the data that doesn't have normal distribution). The quantitative data, such as sex, will be analyzed by using percentage and 95% confident interval for the prevalence.
2. In comparison between two groups, the quantitative data, such as liver fibrosis: positive or negative, will be compared by using t-test (normality) or Mann-Whitney U-test (non-normality) and the quantitative data will be analyzed by Chi-square test or Fisher's exact test. If the results show statistically significance (P-value <0.05) more than one value, the Logistic Regression Analysis will be performed and presented by odds ratio and 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed thalassemia major, for example homozygous beta thalassemia or beta thalassemia/hemoglobin E disease or thalassemia intermedia such as hemoglobin H disease or homozygous Hb CS
2. Age equal to or more than 18 years
3. Previous history of blood transfusion

Exclusion Criteria:

1. Patients who have hepatocellular carcinoma, ascites or pregnancy will be excluded from the study due to the limitation of result interpretation.
2. Unwilling to participate
3. Patient who receiving or completed treatment of hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are thalassemia patients who regularly visit Hematology Clinic, Department of Medicine, Faculty of Medicine Siriraj Hospital
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence and genotypes of HCV infection in thalassemia major and thalassemia intermediate patients who have received blood transfusion in the Department of Medicine, Faculty of Medicine Siriraj Hospital | 1 year

SECONDARY OUTCOMES:
Effect of HCV infection and the risk factors of advanced liver disease and liver cirrhosis in thalassemia major and thalassemia intermediate patients who have received blood transfusion | 1 year
Role of serum HA level and fibrotest in the prediction of cirrhosis in thalassemia major and thalassemia intermediate patients who have received blood transfusion in the Department of Medicine, Faculty of Medicine Siriraj Hospital. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tawesak Tanwandee, Assoc.Prof., Principal Investigator — Division of Gastroenterology, Faculty of Medicine, Siriraj hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Due to patients confidentiality in study protocol. The individual level data will not be released.

REFERENCES:
- [Background] Borgna-Pignatti C, Garani MC, Forni GL, Cappellini MD, Cassinerio E, Fidone C, Spadola V, Maggio A, Restivo Pantalone G, Piga A, Longo F, Gamberini MR, Ricchi P, Costantini S, D'Ascola D, Cianciulli P, Lai ME, Carta MP, Ciancio A, Cavalli P, Putti MC, Barella S, Amendola G, Campisi S, Capra M, Caruso V, Colletta G, Volpato S. Hepatocellular carcinoma in thalassaemia: an update of the Italian Registry. Br J Haematol. 2014 Oct;167(1):121-6. doi: 10.1111/bjh.13009. Epub 2014 Jul 3. PMID 24992281
- [Background] Kountouras D, Tsagarakis NJ, Fatourou E, Dalagiorgos E, Chrysanthos N, Berdoussi H, Vgontza N, Karagiorga M, Lagiandreou A, Kaligeros K, Voskaridou E, Roussou P, Diamanti-Kandarakis E, Koskinas J. Liver disease in adult transfusion-dependent beta-thalassaemic patients: investigating the role of iron overload and chronic HCV infection. Liver Int. 2013 Mar;33(3):420-7. doi: 10.1111/liv.12095. PMID 23402611
- [Background] Wilder J, Patel K. The clinical utility of FibroScan((R)) as a noninvasive diagnostic test for liver disease. Med Devices (Auckl). 2014 May 3;7:107-14. doi: 10.2147/MDER.S46943. eCollection 2014. PMID 24833926
- [Background] Fraquelli M, Cassinerio E, Roghi A, Rigamonti C, Casazza G, Colombo M, Massironi S, Conte D, Cappellini MD. Transient elastography in the assessment of liver fibrosis in adult thalassemia patients. Am J Hematol. 2010 Aug;85(8):564-8. doi: 10.1002/ajh.21752. PMID 20658587
- [Background] Fucharoen S, Winichagoon P. Haemoglobinopathies in southeast Asia. Indian J Med Res. 2011 Oct;134(4):498-506. PMID 22089614
- [Result] Wanachiwanawin W, Luengrojanakul P, Sirangkapracha P, Leowattana W, Fucharoen S. Prevalence and clinical significance of hepatitis C virus infection in Thai patients with thalassemia. Int J Hematol. 2003 Nov;78(4):374-8. doi: 10.1007/BF02983565. PMID 14686498
- [Result] Papastamataki M, Delaporta P, Premetis E, Kattamis A, Ladis V, Papassotiriou I. Evaluation of liver fibrosis in patients with thalassemia: the important role of hyaluronic acid. Blood Cells Mol Dis. 2010 Oct 15;45(3):215-8. doi: 10.1016/j.bcmd.2010.06.002. Epub 2010 Jul 6. PMID 20605573
- [Result] El-Shabrawi MH, Zein El Abedin MY, Omar N, Kamal NM, Elmakarem SA, Khattab S, El-Sayed HM, El-Hennawy A, Ali AS. Predictive accuracy of serum hyaluronic acid as a non-invasive marker of fibrosis in a cohort of multi-transfused Egyptian children with beta-thalassaemia major. Arab J Gastroenterol. 2012 Jun;13(2):45-8. doi: 10.1016/j.ajg.2012.06.006. Epub 2012 Jul 11. PMID 22980590